CLINICAL TRIAL: NCT07077057
Title: Ticino Artificial InTelligence integrAtioN for Occlusion Myocardial Infarction
Acronym: TITAN-OMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Marco Valgimigli, Deputy Chief of Cardiology, Cardiocentro Ticino
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2024-01655
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction (MI); Acute Coronary Syndrome (ACS)
Keywords: Occlusion Myocardial Infarction; Electrocardiogram; Artificial Intelligence
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted ECG interpretation (Experimental): Participants will receive ECG interpretation supported by a CE-marked artificial intelligence (AI) tool (PMcardio, Powerful Medical). The AI output is made available to clinicians in real time, prior to diagnostic or therapeutic decisions, to facilitate earlier identification of occlusion myocardial infarction (OMI) and potentially expedite intervention.
  Interventions: Diagnostic Test: AI-assisted ECG interpretation (PMcardio)
- Standard of Care (No Intervention): Participants will receive standard ECG interpretation without AI support. Clinical decisions regarding diagnosis and treatment will follow usual care pathways, without influence from the AI tool. This arm serves as the comparator to evaluate the added value of AI integration.

INTERVENTIONS:
Diagnostic Test: AI-assisted ECG interpretation (PMcardio) — Participants in the experimental arm will undergo 12-lead ECG interpretation supported by a CE-marked artificial intelligence (AI) tool (PMcardio, Powerful Medical, Slovakia). The AI algorithm analyzes ECG data in real time to detect patterns suggestive of occlusion myocardial infarction (OMI), including cases not meeting traditional ST-elevation myocardial infarction (STEMI) criteria. In the experimental arm, the AI output is provided immediately to the treating clinician and used as an adjunct to standard ECG interpretation to support timely diagnosis and management decisions.
  Arms: AI-assisted ECG interpretation

SUMMARY:
The goal of this clinical trial is to evaluate whether an artificial intelligence (AI)-based ECG interpretation tool improves the early diagnosis and treatment of occlusion myocardial infarction (OMI) in adults presenting with suspected acute coronary syndrome (ACS) who do not meet traditional ST-elevation myocardial infarction (STEMI) criteria.

The main questions it aims to answer are:

1. Does AI-assisted ECG interpretation enable more timely identification and treatment of OMI, as defined by earlier initiation of coronary intervention?
2. Does AI-assisted diagnosis reduce infarct size, measured by peak high-sensitivity troponin T (hsTnT) levels?

Researchers will compare AI-assisted ECG interpretation to standard care to determine if the AI tool improves clinical outcomes and care timelines.

Participants will:

1. Present with symptoms suggestive of ACS but without clear STEMI criteria
2. Be randomized 1:1 to either AI-assisted or standard ECG interpretation
3. Undergo follow-up assessments for cardiovascular outcomes, including 30-day death, time to treatment of total coronary occlusion, and peak hsTnT levels

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms suspected of ongoing acute myocardial ischemia: Patients presenting with symptoms such as chest pain, dyspnoea, sweating, nausea or vomiting, pain radiating to the shoulder/arm/jaw/back, fatigue, or light-headedness
2. Age: Patients aged 18 years or older.
3. Informed Consent: Patients able to provide informed consent

Exclusion Criteria:

1. Clear diagnosis of ST-segment elevation MI (STEMI) according to managing physicians.
2. Pregnancy or Lactation.
3. Legally incompetent to provide informed consent.
4. Symptoms onset>24 hrs prior to clinical presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Hierarchical primary endpoint | 30 days
  The primary endpoint of the prospective phase, analysed hierarchically using the unmatched, unstratified win ratio, will be a composite of:
  * Cardiovascular mortality at 30 days.
  * Timely treatment of angiographically confirmed TIMI 0-1 occlusions, defined as insertion of the arterial sheath within 120 minutes from randomization.
  * Time-to-treatment of angiographically confirmed TIMI 0-1 occlusions.
  * Peak high- hsTnT levels in ng/mL as a surrogate measure of infarct size. Time of coronary intervention will be defined as time from randomisation to insertion of the arterial sheath. Peak hsTnT is defined as the maximum level of hsTnT within 48h from randomization or within 48 hours from intervention if percutaneous coronary intervention took place later than 24 hours from randomization.

SECONDARY OUTCOMES:
Cardiovascular mortality at 30 days | 30 days
  Cardiovascular mortality at 30 days
Timely treatment of TIMI 0-1 occlusions | Periprocedural
  Timely treatment is defined as arterial sheath insertion within 120 minutes of randomization
Time-to-treatment of TIMI 0-1 occlusions | Periprocedural
  Expressed in minutes from time of randomization
Peak hsTnT levels | 48 hours from randomization or intervention
  Peak hsTnT is defined as the maximum level of hsTnT within 48h from randomization or within 48 hours from intervention if percutaneous coronary intervention took place later than 24 hours from randomization.
Major adverse cardiovascular events (MACE) at follow-up | up to 10 years
  Major adverse cardiovascular events (MACE), defined as a composite of cardiovascular death, myocardial infarction, or stroke at follow up (30-days, 1 year, 3/5/10 years)
Cardiovascular death at follow-up | up to 10 years
  Cardiovascular death at follow up (30-days, 1 year, 3/5/10 years)
Myocardial infarction at follow-up | up to 10 years
  Myocardial infarction at follow up (30-days, 1 year, 3/5/10 years)
Stroke at follow-up | up to 10 years
  Stroke at follow up (30-days, 1 year, 3/5/10 years)
Infarct Size | 48 hours from randomization or intervention
  • hsTnT area under the curve
Infarct Size | 48 hours from randomization or intervention
  • Creatine kinase-MB (CK-MB) peak concentration
Infarct Size | 48 hours from randomization or intervention
  • CK-MB area under the curve
Time from randomization to antithrombotic therapy | periprocedural
  Time from randomization to antithrombotic therapy (expressed in minutes)
Time from randomization to coronary angiography | periprocedural
  Time from randomization to coronary angiography (expressed in minutes) This outcome will be assessed both in all patients and in patients with OMI according to the different definitions.
Angiographic outcomes (restricted to patients undergoing PCI) | Periprocedural
  * Worst TIMI flow grade post-PCI (0-3)
  * Worst TIMI thrombus grade post-PCI (0-5)
Total time spent in the emergency department post-randomization | periprocedural
  Total time spent in the emergency department post-randomization
Length of hospital stay post-randomization | up to 30 days
  Length of hospital stay post-randomization (days)
Resource utilization | periprocedural
  Number of diagnostic tests and procedures performed post-randomization before coronary angiography, including troponin measurements, transthoracic echocardiography and stress testing
Health economic outcomes | 30 days
  These include both direct and indirect costs.
  Direct costs are defined as medical costs incurred post-randomization during the index hospitalization or emergency department visit, including diagnostics and procedures (e.g., ECG, troponin testing, coronary angiography, PCI), medications and consumables, staff time, and length of stay.
  Indirect costs, defined as non-medical or societal costs up to 30 days post-randomization, including lost productivity (e.g., time off work for patients or caregivers), transportation to follow-up visits, informal caregiving support, and early rehabilitation services
Safety (Serious adverse events) | up to 10 years
Diagnostic accuracy of AI algorithm | periprocedural
  Restricted to patients in the control group:
  * Sensitivity
  * Specificity
  * Positive predictive value (PPV)
  * Negative predictive value (NPV)
Quality of life (EQ-5D-5L) | up to 30 days
  Health-related quality of life, assessed using the EQ-5D-5L instrument at discharge and 30 days post-randomization

OTHER OUTCOMES:
Pre-procedural ECG analysis | periprocedural
  Sensitivity analysis of diagnostic accuracy of the AI-algorithm based on the 12-lead ECG recorded immediately prior to the start of coronary angiography, instead of the ECG at presentation.
Alternative OMI definitions | 30 days
  Sensitivity analysis of the primary outcome using an alternative definition of OMI: TIMI flow 0-1, or TIMI flow 2-3 in the presence of large thrombus burden (TIMI thrombus grade ≥3).

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocentro Ticino Institute, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: Reasonable request